CLINICAL TRIAL: NCT03423680
Title: A Multicenter, Randomized, Double Blind, Placebo-controlled, Parallel Group, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of Abilify® Tablet(Aripiprazole) as an Adjunctive Treatment in the Treatment of Major Depressive Episode Associated With Bipolar I or II Disorder
Brief Title: A Study of Abilify® Tablet(Aripiprazole) as an Adjunctive Treatment in the Bipolar Depression
Acronym: APOLLO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 031-402-00154
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abilify (Tablet) (Experimental)
  Interventions: Drug: Abilify 2, 5, 10, 15mg (Tablet)
- Placebo of Abilify (Tablet) (Placebo Comparator)
  Interventions: Drug: Placebo of Abilify 2, 5, 10, 15mg (Tablet)

INTERVENTIONS:
Drug: Abilify 2, 5, 10, 15mg (Tablet) — Randomized subjects will take 1 tablet of aripiprazole or placebo orally once daily from the baseline visit (Visit 2) to Visit 8 (Week 8 visit or discontinuation visit). The initial dose of aripiprazole, the investigational product, is 2 mg once daily (irrespective of meals), which the investigators can maintain, increase or decrease within a range of 2 - 15 mg at each scheduled study visit, depending on the subject's clinical response and tolerability.
  Arms: Abilify (Tablet)
Drug: Placebo of Abilify 2, 5, 10, 15mg (Tablet) — Randomized subjects will take 1 tablet of aripiprazole or placebo orally once daily from the baseline visit (Visit 2) to Visit 8 (Week 8 visit or discontinuation visit). The initial dose of aripiprazole, the investigational product, is 2 mg once daily (irrespective of meals), which the investigators can maintain, increase or decrease within a range of 2 - 15 mg at each scheduled study visit, depending on the subject's clinical response and tolerability.
  Arms: Placebo of Abilify (Tablet)

SUMMARY:
This is an 8-week, multicenter, randomized, double blind, placebo controlled study to evaluate the efficacy and safety of aripiprazole as an adjunctive treatment with mood stabilizer for the treatment of patients (outpatients or inpatients) with type I or II bipolar disorder accompanied by major depressive episode, without any psychotropic features.

This study involves patients who are considered by the investigator not to have a proper improvement, despite receiving a mood stabilizer (lithium or valproic acid) for a sufficient (≥ 28 days) period of time during the current depressive episode.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 19 and < 70 years at the time of informed consent
* Patients who are able to understand information required for providing a consent
* Patients who have received a mood stabilizer (lithium or valproic acid)
* Patients with bipolar I or II disorder accompanied by major depressive episode
* Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥ 20 at both the screening and baseline visits

Exclusion Criteria:

* Patients diagnosed with bipolar I or II disorder with mania, mixed or psychotropic features
* Patients considered to have a high risk of suicide during the study period by the investigator based on current psychotic symptom and the patient's past medical history

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in the Montgomery-Åsberg Depression Rating Scale total score | Week 8
  Mean change in the MADRS total score from baseline to the end of the study(Week 8) The total score ranges from 0 to 60. Higher score indicates more severe depression.

SECONDARY OUTCOMES:
Mean change in the Clinical Global Impression-BP version Severity of Illness (Depression) score | Week 8
  The score ranges from 1 to 7. Higher score indicates more severe depression.
Response rate | Week 8
Remission rate | Week 8
Percentage of subjects with Clinical Global Impression-BP version Severity of Illness (Depression) score of 1 or 2 | Week 8
  The score ranges from 1 to 7. Higher score indicates more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Seounl National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No